CLINICAL TRIAL: NCT03890523
Title: Covered Metallic Segmented Airway Stent Modified With 3D Printing for Gastro-respiratory Fistula Involving Carina and Distal Bronchi
Brief Title: Airway Stent Modified With 3D Printing for Gastro-respiratory Fistula Involving Carina and Distal Bronchi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other); Shanghai Tong Ren Hospital (Other); Ruijin Hospital Luwan Branch (Other)
Responsible Party: Principal Investigator, Zhongmin Wang, Principal Investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: airwaystentfistula
Record Dates: First submitted 2019-03-19; First posted 2019-03-26 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Airway Disease; Fistula Bronchial; Fistula, Gastric
Keywords: 3D printed; airway stent; carina; distal bronchi
MeSH Terms: conditions — Bronchial Fistula; Gastric Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Segmented Airway Stent for Gastro-Respiratory fistula (Experimental): Segmented covered metallic airway stent modified with 3D printing was used for gastro-respiratory fistula.
  Interventions: Procedure: Airway stent implantation

INTERVENTIONS:
Procedure: Airway stent implantation — The segmented airway stent modified with 3D printing were implanted to treat gastro-respiratory fistula involving carina and distal bronchi. The stents were removed because of stent-related complications or tracheobronchial healing.
  Other Names: Stent removal

SUMMARY:
In this study, the investigators used the covered metallic segmented airway stent modified with 3D printing to treat gastro-respiratory fistula involving carina and distal bronchi and aimed to determine the feasibility, efficacy and safety of this technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastro-respiratory fistula involving carina and bronchi distal to carina based on the diagnosis by bronchoscopy , gastroscopy and CT.
* The patients who could not tolerate surgery and did not have clinical improvement after conservative treatment.

Exclusion Criteria:

* Severe infection
* coagulation disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Relief of symptoms | 1 month
  Main symptoms as follows: cough, dysphagia, dyspnea, and expectoration.
Heal of fistula | 3 months
  The heal of fistula confirmed by gastroscopy, bronchoscopy and CT

SECONDARY OUTCOMES:
Number of participants with adverse events that are related to stent implantation | 6 months
  Adverse events as follows: migration of the stent, severe chest pain, hemoptysis, granuloma formation, pneumonia and accumulation of secretion
Stent patency time | 6 months
  Stent patency time is defined as the time from the stent implantation to stent restenosis or death due to any cause, or censored at date last known alive

CONTACTS AND LOCATIONS:
Overall Officials: Zhongmin Wang, MD, Principal Investigator — Ruijin Hospital
Locations (2):
- China (2):
  - Shanghai Tongren Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital Luwan Branch, Shanghai

IPD SHARING:
Plan to Share IPD: No